CLINICAL TRIAL: NCT04848883
Title: Infectious Diseases Experts as Part of the Antibiotic Stewardship Team in Primary Care: Protocol for a Cluster-randomised Blinded Study (IDASP)
Brief Title: Infectious Diseases Experts as Part of the Antibiotic Stewardship Team in Primary Care
Acronym: IDASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Ariadna Padullés Zamora, Principal Investigator, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PR277/19
Record Dates: First submitted 2021-03-22; First posted 2021-04-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Infectious Disease
Keywords: Antimicrobial stewardship program; Primary care; Infectious disease specialist; Bacterial resistance
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Six primary care centres will be randomised by conglomerates in 3 parallel groups. First group with three randomised centres will receive a conventional AMS, meanwhile the three other parallel randomised centres will include an infectious diseases specialist in the AMS group and a biweekly meetings.
  List of study sites: El Castells from Castelldefels, Prat de Llobregat 2, Gava 1, Viladecans 2, Hospitalet de Llobregat 2 Sant Josep and Santa Eulàlia Nord.
Who Masked: Outcomes Assessor
Masking Description: Evaluators of secondary outcomes will be blind related to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced AMS program (Experimental): Three randomily assigned primary care centres in which an infectious diseases expert will be continuously in touch with primary care practitioners.
  Interventions: Behavioral: Advanced AMS program; Behavioral: Standard AMS program
- Standard AMS program (Active Comparator): Three primary care centres in which a typical AMS will be promoted.
  Interventions: Behavioral: Standard AMS program

INTERVENTIONS:
Behavioral: Advanced AMS program — 1. - Telephone acces to infectious disease experts to discuss patients' therpies during working days.
  2. - Biweeckly meetings with infectious diseases experts and antimicrobial stewardship group.
  Arms: Advanced AMS program
Behavioral: Standard AMS program — 1. - Educational materials.
  2. - Updated local antibiotic guidelines.
  3. - Promotion of delayed antibiotic prescription.
  4. - Promotion of Streptococcus pyogenes antigen test (Streptotest) if bacterial tonsillitis is suspected.
  5. - Daily report to GP of multiresistant bacteria isolates in urinary samples.
  6. - Quarterly reports to prescribers of AMS outcomes at the centre-level.

SUMMARY:
A cluster-randomised multicentre blinded clinical trial will be performed in six primary care centres located in the southern metropolitan area of Barcelona (Spain). The objective is to assess whether including experts on infectious diseases (ID) within the antimicrobial stewardship (AMS) team of primary care achieves higher reductions on overall antibiotic consumption and increases the quality of prescription in diagnosed upper respiratory and urinary tract infections.

Centres will be randomly assigned to receive a standard-AMS or an advanced-AMS (intervention). Advanced-AMS includes all standard-AMS strategies plus general practitioner chance to discuss clinical cases by telephone to ID expert on working days (8:00 am to 8:00 pm), and by biweekly meetings.

DETAILED DESCRIPTION:
STUDY DESIGN. A cluster-randomised, multicentre blinded clinical trial will be conducted in six primary care centres between June 2021 and June 2023.

This cluster-randomised trial uses primary care centres as a unit of analysis to avoid intracentre contamination.

SCOPE OF STUDY. Six primary care centres in the southern metropolitan area of Barcelona.

SUBJECTS OF STUDY. General practitioners of the participating centres. Paediatricians are excluded. Patients older than 14 years who have a diagnosis of upper respiratory tract or urinary tract infections will be prospectively follow up to assess information related to secondary outcomes. Each patient could be included more than once if the GP visit is 30 days or more apart from the initial medical assessment.

Eligible patients will be identified following the International Classification of Diseases (ICD-10) CM codes as follows:

Upper respiratory tract infection: J00, J01, J02, J03, J04, J05, J06, J31, J39, H60, H62, H65, H66, H67, H83 and H92.

Urinary tract infection: N10, N30, N39, N41, R82 and O23.

TIMELINE. From June to September 2021 standard-AMS will be promoted to increase understanding and acceptance of AMS by general practitioners. Baseline data collection will begin on October 2021 and will last six months. After these six months, on 1 April 2022, centres will be randomly assigned to receive an advanced-AMS, or to continue the standard-AMS. The intervention will be spanned 12 months, until 31 March 2023.

RANDOMISATION. A centralised electronic computer system will generate a random list based on permuted blocks. To ensure similar characteristics among centres permuted blocks will be created with stratification on the total number of referral population and the number of population older than 65 years old by centre. Investigators will be unaware of the block size and the permutation procedure.

STUDY GROUPS. The 6 centres will be assigned to receive an advanced AMS or a standard AMS, 3 in one and 3 in another. The standard AMS will receive an standard antibiotic optimization program based on:

1. Educational campaign addressed both, to patients and health professionals, to increase awareness about antibiotic indications and potential harms of its misuse.
2. Updated local antibiotic empirical guidelines for treating common infections according to local resistance patterns.
3. Promotion of delayed antibiotic prescription.
4. Promotion of Streptococcal pyogenes antigen test (Streptotest) if bacterial tonsillitis is suspected.
5. Daily microbiological report of resistant bacteria isolates to general practitioners.
6. Annual reports to prescribers of main AMS outcomes at centre-level.

The advanced AMS group will have the same standard AMS program, enhanced with:

* Telephone access to ID expert on working days (8:00 am to 8:00 pm).
* Biweekly meetings among GP and infectious diseases experts to discuss clinical cases.

More detailed data are placed forward in the document.

BLINDING. Two secondary end-points (unnecessary antibiotic therapy and adequacy of therapy), will be evaluated by two independent investigators who will be blinded to centre allocation. Discrepant decisions among them will be discussed with a third blinded physician to achieve consensus. The degree of agreement will be recorded with the kappa statistic analysis. The centre allocation will not be blinded for the participating centres and general practitioners.

OUTCOMES. Outcomes will be measured in each primary centre with a mensual periodicity during 12 consecutive months. These variables are:

* Main objective. To assess the impact of advanced-AMS on overall antibiotic consumption measured by defined daily dose of antibiotic per 1.000 inhabitants per day (DHD).
* Secondary objectives:

  * To assess the impact of the advanced-AMS on unnecessary antibiotic prescriptions in diagnosed upper respiratory and urinary tract infections.
  * To evaluate the impact of the advanced-AMS on the adequacy of antibiotic prescriptions.
  * To evaluate the impact of the advanced-AMS on the total number of re-attendance to general practitioners or emergency department for any reason within 30 days after the initial GP evaluation.
  * To evaluate the impact of the advanced-AMS on the number of hospital admissions for any reason within 30 days after the initial GP visit.

DEFINITIONS.

* DHD are calculated by the following the World Health Organisation criteria (https://www.who.int/tools/atc-ddd-toolkit/indicators).
* Unnecessary prescription will be considered as follows:

  * An antibiotic prescribed in upper respiratory infections, which is in disagreement with the local antibiotic guidelines.
  * An antibiotic is prescribed in asymptomatic bacteriuria, which is defined as having a positive urine culture with ≥ 10EXP5 CFU/ml of an uropathogen in patients without signs or symptoms of urinary tract infection (dysuria, urinary frequency or urgency, suprapubic pain, fevers, or flank pain). Pregnant women and patients undergoing urologic interventions are excluded from this definition.
* Adequacy of antibiotic therapy will be considered when prescription fulfils the local guidelines: type of antibiotic + dose, and length of therapy.

DATA COLLECTION AND MONITORING. Monthly DHD will be calculated based on the dispensing data of our electronic prescribing system of the Catalan Institute of Health.

To get information regarding secondary outcomes, patients who fulfil ICD-10 CM codes on the last working day of every month will be selected by a cross-sectional analysis. On these selected patients, information from electronic medical records (SAP logon® and eCAP) will be obtained. Investigator will obtain the following variables: demographics, Charlson score, type of infection, antibiotic prescribed, doses and length of antibiotic therapy, re-attendance to the general practitioner, attendance to the emergency department, and hospital admission. All the included patients will be followed up 30 days after the initial primary care physician visit. To ensure completeness of data, a telephone call will be allowed if any crucial data is missing in the electronic medical record.

Information regarding the burden of the intervention such as the number of telephone calls received by the ID expert per month and the number of participants to biweekly meetings with the ID will be also collected.

All data will be recorded by the study monitor on a standardized data abstraction form by using RedCap (Research Electronic Data Capture) hosted at IDIBELL, a secure web application for building and managing online databases.

SAMPLE SIZE. The intervention area has a total of 18 primary care centres and a reference population of 402 657 inhabitants. Six centres will be included, three in each study arm, implying an approximate coverage of 37% of the referral population (147 644 inhabitants). The consumption of antibiotics in 2017 was 8.94 DHD, and it's expected to reduce this consumption by 10% in the intervention group. The number of 3 clusters per arm will allow rejecting the null hypothesis of equal consumption with a power of 80%, assuming a moderate intra-cluster correlation of 0.2, an intra-cluster variance of 4, and a mean difference of 1 DHD. Type I error is set at 5%.

STATISTICAL ANALYSIS. A descriptive analysis will be performed on the monthly consumption of antibiotics expressed in DHD by the study group (control and intervention), period, and cluster. The monthly consumption of antibiotics evolution will be represented on a graph by months, and a smoothed curve will be estimated using locally weighted smoothing (LOESS).

Antibiotic consumptions will be compared according to the study group using a time series model. Where the dependent variable will be the monthly consumption of antibiotics expressed in DHDs and the independent variable will be the study group. In the estimation of the model, the seasonality, the trend, and the first and second-order lags of the series will be analyzed. Also, the use of hierarchical models due to cluster design will be taken into account.

A descriptive analysis of the demographic and clinical profile of the patients surveyed will be performed. A McNemar test will be used to compare, between the study groups, the percentage of patients with an unnecessary prescription for the upper respiratory and urinary tract, the percentage of patients with an adequate prescription according to the guidelines, the percentage of patients who revisit general practitioner or emergency room at 30 days, and the percentage of patients with hospital admission at 30 days. Also, log-binomial regression models will be performed, to estimate the effect of the intervention in terms of risk on the above-mentioned outcomes adjusting by patients' clinical profile. To estimate models it will be accounted that patients are nested in primary care clusters, so a correction of the standard errors is carried out through the variance-covariance matrix.

Data management and statistical analysis will be carried out with the statistical package R version 4.0.1 or higher.

LIMITATIONS. The study does not contemplate randomisation by prescribing physician, but by conglomerates to avoid possible contamination effects at the prescribing physician and patients in the same centre. As it is a cluster analysis, there could be differences in the degree of prescription of doctors within the same centre and between the different centres. In order to reduce this problem, the variability of prescribing intra-cluster and between clusters has been calculated during the period 2017 in a group of primary care centres in the intervention area, differences that have been taken into account for the calculation of the sample. Design of the present study does not include a third group without any AMS intervention due to department policies during 2019. However, to achieve the best result interpretation, an historic of the antibiotic consumption in the participating centres will act as a control group, and a baseline period with only an standard-AMS intervention will be performed.

Comparisons between all stages of the clinical trial will be performed to obtain more robust data.

ETHICAL ASPECTS. This research will be carried out under the standards of good clinical practices following the principles of the Declaration of Helsinki (Fortaleza, 2013), as well as the current legislation applicable to this type of study. This study has been approved by the Ethics Committee of Hospital Universitari de Bellvitge and the Foundation University Institute for Primary Health Care Research Jordi Gol i Gurina (IDIAPJGol) who waived the need to obtain informed consent since the intervention is mainly aimed at health-care professionals (general practitioners) who will be previously informed of the objective and other relevant aspects of the study (REF. PR277/19 - REF. 4R20/26).

Clinical data treatment of the included patients in the research project as well as that of associated professionals (primary care physicians) will be carried out following the established by the Organic Law 3/2018, of December 5, and by Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016 on Data Protection (RGPD). Based on these regulations, the sponsor will guarantee the protection of the confidentiality of the participants in the program, both patients and doctors.

The data collection sheets will be identified with a code. The name of the doctor or patient will not appear in any document, or any publication or communication of the study results.

ELIGIBILITY:
All general practitioners of the 6 primary care centers will be included in our clinical trial, excepting paediatricians. Data collection will be performed on patients attended in these centres. Inclusion and exclusion criteria will be applied on the patients attended by general practitioners:

Inclusion criteria:

* Patients older than 14 years old diagnosed with respiratory infections: pharyngoamygdalitis, sinusitis and otitis.
* Patients older than 14 years old diagnosed with urinary tract infections: cystitis, prostatitis and pyelonephritis.

Exclusion criteria:

* Patients less than 14 years old.
* Patients with indwelling urinary catheter.
* Patients with congenital urinary tract abnormalities.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
To asses the impact of implementing an advanced-AMS program (inclusion of infectious diseases specialists) on the overall antibiotic consumption. | Through study completion, an average of 1 year and a half
  Antibiotic defined daily dose per 1,000 inhabitant's day (DHD).

SECONDARY OUTCOMES:
Number of patients with unnecessary antibiotic prescriptions on high respiratory pathway infections. | Through study completion, an average of 1 year and a half
  Analysis of all patients attended in primary care centers with high respiratory tract infections. Unnecessary antibiotic prescription will be all those prescriptions which are in disagreement with the local antibiotic guidelines.
Number of patients with unnecessary antibiotic prescriptions on urinary tract infections. | Through study completion, an average of 1 year and a half
  Checking all patients attended in primary care centers with urinary tract infections. Unnecessary antibiotic prescription will be all those prescriptions which are in disagreement with the local antibiotic guidelines.
Number of patients with an adequate antibiotic treatment | Through study completion, an average of 1 year and a half
  Checking antibiotic treatment of all patients attended in primary care centers with both urinary and respiratory tract infection. Adequation will be determined by two different blinding investigators who will receive the information of type of antibiotic, dose and length of treatment. Discrepant decisions among them will be discussed with a third blinded physician.
Number of patients re-consulting after completing antibiotic therapy. | Through study completion, an average of 1 year and a half
  Checking any type of re-consulting of all patients attended in primary care centers with both urinary and respiratory tract infection after completing antibiotic treatment, during 30 days after the patients consult with the general practitioner.
Number of cases who needs hospitalisation 30 days after antibiotic therapy. | Through study completion, an average of 1 year and a half
  Checking any type of hospitalisation of all patients attended in primary care centers with both urinary and respiratory tract infection after completing antibiotic treatment, during 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna Padullés, Pharmacyst, Study Director — Institut d'Investigació Biomèdica de Bellvitge; Evelyn Shaw, Doctor, Principal Investigator — Institut d'Investigació Biomèdica de Bellvitge
Locations (1):
- Hospital Univeristari de Bellvitge, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buehrle DJ, Shively NR, Wagener MM, Clancy CJ, Decker BK. Sustained Reductions in Overall and Unnecessary Antibiotic Prescribing at Primary Care Clinics in a Veterans Affairs Healthcare System Following a Multifaceted Stewardship Intervention. Clin Infect Dis. 2020 Nov 5;71(8):e316-e322. doi: 10.1093/cid/ciz1180. PMID 31813965
- [Background] Brinkmann I, Kibuule D. Effectiveness of antibiotic stewardship programmes in primary health care settings in developing countries. Res Social Adm Pharm. 2020 Sep;16(9):1309-1313. doi: 10.1016/j.sapharm.2019.03.008. Epub 2019 Mar 16. PMID 30904409
- [Background] Laxminarayan R, Duse A, Wattal C, Zaidi AK, Wertheim HF, Sumpradit N, Vlieghe E, Hara GL, Gould IM, Goossens H, Greko C, So AD, Bigdeli M, Tomson G, Woodhouse W, Ombaka E, Peralta AQ, Qamar FN, Mir F, Kariuki S, Bhutta ZA, Coates A, Bergstrom R, Wright GD, Brown ED, Cars O. Antibiotic resistance-the need for global solutions. Lancet Infect Dis. 2013 Dec;13(12):1057-98. doi: 10.1016/S1473-3099(13)70318-9. Epub 2013 Nov 17. PMID 24252483
- [Background] Cassini A, Hogberg LD, Plachouras D, Quattrocchi A, Hoxha A, Simonsen GS, Colomb-Cotinat M, Kretzschmar ME, Devleesschauwer B, Cecchini M, Ouakrim DA, Oliveira TC, Struelens MJ, Suetens C, Monnet DL; Burden of AMR Collaborative Group. Attributable deaths and disability-adjusted life-years caused by infections with antibiotic-resistant bacteria in the EU and the European Economic Area in 2015: a population-level modelling analysis. Lancet Infect Dis. 2019 Jan;19(1):56-66. doi: 10.1016/S1473-3099(18)30605-4. Epub 2018 Nov 5. PMID 30409683
- [Background] Dellit TH, Owens RC, McGowan JE Jr, Gerding DN, Weinstein RA, Burke JP, Huskins WC, Paterson DL, Fishman NO, Carpenter CF, Brennan PJ, Billeter M, Hooton TM; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America. Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America guidelines for developing an institutional program to enhance antimicrobial stewardship. Clin Infect Dis. 2007 Jan 15;44(2):159-77. doi: 10.1086/510393. Epub 2006 Dec 13. No abstract available. PMID 17173212
- [Background] Rodriguez-Bano J, Pano-Pardo JR, Alvarez-Rocha L, Asensio A, Calbo E, Cercenado E, Cisneros JM, Cobo J, Delgado O, Garnacho-Montero J, Grau S, Horcajada JP, Hornero A, Murillas-Angoiti J, Oliver A, Padilla B, Pasquau J, Pujol M, Ruiz-Garbajosa P, San Juan R, Sierra R; Grupo de Estudio de la Infeccion Hospitalaria-Sociedad Espanola de Enfermedades Infecciosas y Microbiologia Clinica; Sociedad Espanola de Farmacia Hospitalaria; Sociedad Espanola de Medicina Preventiva, Salud Publica e Higiene. [Programs for optimizing the use of antibiotics (PROA) in Spanish hospitals: GEIH-SEIMC, SEFH and SEMPSPH consensus document]. Enferm Infecc Microbiol Clin. 2012 Jan;30(1):22.e1-22.e23. doi: 10.1016/j.eimc.2011.09.018. Epub 2011 Dec 15. Spanish. PMID 22178010
- [Background] Fleming-Dutra KE, Hersh AL, Shapiro DJ, Bartoces M, Enns EA, File TM Jr, Finkelstein JA, Gerber JS, Hyun DY, Linder JA, Lynfield R, Margolis DJ, May LS, Merenstein D, Metlay JP, Newland JG, Piccirillo JF, Roberts RM, Sanchez GV, Suda KJ, Thomas A, Woo TM, Zetts RM, Hicks LA. Prevalence of Inappropriate Antibiotic Prescriptions Among US Ambulatory Care Visits, 2010-2011. JAMA. 2016 May 3;315(17):1864-73. doi: 10.1001/jama.2016.4151. PMID 27139059
- [Background] Smieszek T, Pouwels KB, Dolk FCK, Smith DRM, Hopkins S, Sharland M, Hay AD, Moore MV, Robotham JV. Potential for reducing inappropriate antibiotic prescribing in English primary care. J Antimicrob Chemother. 2018 Feb 1;73(suppl_2):ii36-ii43. doi: 10.1093/jac/dkx500. PMID 29490058
- [Background] Dyar OJ, Beovic B, Pulcini C, Tacconelli E, Hulscher M, Cookson B; ESCMID generic competencies working group. ESCMID generic competencies in antimicrobial prescribing and stewardship: towards a European consensus. Clin Microbiol Infect. 2019 Jan;25(1):13-19. doi: 10.1016/j.cmi.2018.09.022. Epub 2018 Nov 8. PMID 30414817
- [Background] Alvarez-Lerma F, Grau S, Echeverria-Esnal D, Martinez-Alonso M, Gracia-Arnillas MP, Horcajada JP, Masclans JR. A Before-and-After Study of the Effectiveness of an Antimicrobial Stewardship Program in Critical Care. Antimicrob Agents Chemother. 2018 Mar 27;62(4):e01825-17. doi: 10.1128/AAC.01825-17. Print 2018 Apr. PMID 29339385
- [Background] Molina J, Penalva G, Gil-Navarro MV, Praena J, Lepe JA, Perez-Moreno MA, Ferrandiz C, Aldabo T, Aguilar M, Olbrich P, Jimenez-Mejias ME, Gascon ML, Amaya-Villar R, Neth O, Rodriguez-Hernandez MJ, Gutierrez-Pizarraya A, Garnacho-Montero J, Montero C, Cano J, Palomino J, Valencia R, Alvarez R, Cordero E, Herrero M, Cisneros JM; PRIOAM team. Long-Term Impact of an Educational Antimicrobial Stewardship Program on Hospital-Acquired Candidemia and Multidrug-Resistant Bloodstream Infections: A Quasi-Experimental Study of Interrupted Time-Series Analysis. Clin Infect Dis. 2017 Nov 29;65(12):1992-1999. doi: 10.1093/cid/cix692. PMID 29020166
- [Background] Roca I, Akova M, Baquero F, Carlet J, Cavaleri M, Coenen S, Cohen J, Findlay D, Gyssens I, Heuer OE, Kahlmeter G, Kruse H, Laxminarayan R, Liebana E, Lopez-Cerero L, MacGowan A, Martins M, Rodriguez-Bano J, Rolain JM, Segovia C, Sigauque B, Tacconelli E, Wellington E, Vila J. The global threat of antimicrobial resistance: science for intervention. New Microbes New Infect. 2015 Apr 16;6:22-9. doi: 10.1016/j.nmni.2015.02.007. eCollection 2015 Jul. PMID 26029375
- [Background] Castro-Sanchez E, Moore LS, Husson F, Holmes AH. What are the factors driving antimicrobial resistance? Perspectives from a public event in London, England. BMC Infect Dis. 2016 Sep 2;16(1):465. doi: 10.1186/s12879-016-1810-x. PMID 27590053
- [Background] Bell BG, Schellevis F, Stobberingh E, Goossens H, Pringle M. A systematic review and meta-analysis of the effects of antibiotic consumption on antibiotic resistance. BMC Infect Dis. 2014 Jan 9;14:13. doi: 10.1186/1471-2334-14-13. PMID 24405683
- [Background] MacDougall C, Polk RE. Antimicrobial stewardship programs in health care systems. Clin Microbiol Rev. 2005 Oct;18(4):638-56. doi: 10.1128/CMR.18.4.638-656.2005. PMID 16223951
- [Background] Steinman MA, Landefeld CS, Gonzales R. Predictors of broad-spectrum antibiotic prescribing for acute respiratory tract infections in adult primary care. JAMA. 2003 Feb 12;289(6):719-25. doi: 10.1001/jama.289.6.719. PMID 12585950
- [Background] Llor C, Moragas A, Hernandez S, Crispi S, Cots JM. Misconceptions of Spanish general practitioners' attitudes toward the management of urinary tract infections and asymptomatic bacteriuria: an internet-based questionnaire study. Rev Esp Quimioter. 2017 Oct;30(5):372-378. Epub 2017 Jul 24. PMID 28737026
- [Background] Rousham E, Cooper M, Petherick E, Saukko P, Oppenheim B. Overprescribing antibiotics for asymptomatic bacteriuria in older adults: a case series review of admissions in two UK hospitals. Antimicrob Resist Infect Control. 2019 May 2;8:71. doi: 10.1186/s13756-019-0519-1. eCollection 2019. PMID 31073402
- [Background] Nicolle LE, Gupta K, Bradley SF, Colgan R, DeMuri GP, Drekonja D, Eckert LO, Geerlings SE, Koves B, Hooton TM, Juthani-Mehta M, Knight SL, Saint S, Schaeffer AJ, Trautner B, Wullt B, Siemieniuk R. Clinical Practice Guideline for the Management of Asymptomatic Bacteriuria: 2019 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2019 May 2;68(10):e83-e110. doi: 10.1093/cid/ciy1121. PMID 30895288
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Derived] Ronda M, Padulles A, Simonet P, Rodriguez G, Estrada C, Lerida A, Ferro JJ, Cobo S, Tubau F, Gardenes L, Freixedas R, Lopez M, Carrera E, Pallares N, Tebe C, Carratala J, Puig-Asensio M, Shaw E. Infectious diseases experts as part of the antibiotic stewardship team in primary care: protocol for a cluster-randomised blinded study (IDASP). BMJ Open. 2021 Oct 11;11(10):e053160. doi: 10.1136/bmjopen-2021-053160. PMID 34635529